CLINICAL TRIAL: NCT03792386
Title: Clinical Visibility of Combined Ultrasound and Fluoroscopy Guided Cervical Transforaminal Injection
Brief Title: Combined Ultrasound and Fluoroscopy Guided Cervical Transforaminal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R/17.06.52
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Chronic Cervical Radicular Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guidance with fluoroscopic confirmation (Active Comparator): Patients in which the intervention will be performed using ultrasound guidance with fluoroscopic confirmation
  Interventions: Procedure: Ultrasound guidance with fluoroscopic confirmation
- Fluoroscopic guidance with ultrasonographic confirmation. (Active Comparator): Patients in which intervention will be performed using fluoroscopic guidance with ultrasonographic confirmation.
  Interventions: Procedure: Fluoroscopic guidance with ultrasonographic confirmation.

INTERVENTIONS:
Procedure: Ultrasound guidance with fluoroscopic confirmation — the cervical spine will be sonographically examined to determine the C7 transverse process then after lidocaine skin infiltration, a 22G spinal needle is directed towards the hypoechoic shadow of the nerve root using the in-plane technique. then 1ml of non-ionic contrast will be injected and AP and the oblique foraminal fluoroscopic view will be obtained. After confirmation of correct placement of the needle,(2ml, 8mg dexamethasone plus 1ml Lidocaine 1%) will be injected.
  Arms: Ultrasound guidance with fluoroscopic confirmation
Procedure: Fluoroscopic guidance with ultrasonographic confirmation. — After AP view, alignment or squaring of the target lower end plate, an oblique foraminal view is obtained. Following lidocaine 1% skin infiltration, a 22G spinal needle is directed towards the target foramen then, the superficial ultrasound probe will be applied to delineate the foramen. The needle will be advanced ~3mm towards the dorsal root ganglia under fluoroscopic guidance. After contrast confirmation of needle placement, 2ml,8mg dexamethasone plus 1ml Lidocaine 1%) will be injected.
  Arms: Fluoroscopic guidance with ultrasonographic confirmation.

SUMMARY:
The combined use of Doppler ultrasound and fluoroscopy may increase efficacy and safety during cervical transforaminal epidural injection of steroid and local anaesthetic

The study will detect by which technique we have to start and confirm by the other to reach the favourable outcome.

DETAILED DESCRIPTION:
In a previous Ultrasound study involving the C5C6 levels, a performance time of 248.8 ± 82.7 seconds was reported. On the basis of these findings, a 30% difference in performance time would represent an effect size of 0.82 and would require 20 patients per group to achieve an alpha error of 0.05 and beta error of 0.1. For dropped cases; 5% will be added. So a total sample size of 64 patients (32 per group) will be required.

Statistical Analysis: will be performed using SPSS version 22 statistical software. For quantitative data, normality will be first assessed with the Shapiro test and then analyzed with the Student t-test. Data that will not have a normal distribution, as well as ordinal data, will be analyzed with the Mann-Whitney U test. For binomial data, Fisher exact test will be used. All P values presented will be 2-sided and values of less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from radicular discogenic pain
* Patients suffering from radicular foraminal pain Patients suffering from radicular pain secondary to spinal canal stenosis
* Patients suffering from radicular pain after failed cervical disc surgery
* Not responding to conservative management for at least 3 months
* Patients with recalcitrant symptoms after transforaminal steroid injection.
* American Society of Anesthesiology (ASA) from I to III

Exclusion Criteria:

* Presence of local or systemic infection
* Coagulopathy
* Body mass index > 35
* Cervical spine fracture
* Myelopathy
* Malignancy
* Pregnancy
* Patients unable to communicate with the operator during the procedure or report their pain diary after it.
* Patients not responding to previous cervical transforaminal steroid injection or had any untoward effects.
* Allergy to any one of the used medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
performance time in minutes | starting by direction of the spinal needle towards the nerve root till confirmation of correct placement of the needle and injection over a period of 15 minutes
  Defined as time needed for correct transforaminal needle placement through ultrasound guidance followed by fluoroscopic confirmation or fluoroscopic guidance followed by ultrasound confirmation

SECONDARY OUTCOMES:
Feasibility of the radiologic target | starting by direction of the spinal needle towards the nerve root till confirmation of correct placement of the needle and injection over a period of 15 minutes
  number of needle corrections till confirmation of correct placement of the needle
Visual analogue score | pre-procedure then every 3 months till 6 months after the procedure
  Visual analogue score (VAS, 11-point scale): using 100mm visual analogue score in which 0 mm represents no pain and 100mm worst pain imaginable
Neck disability index | pre-procedure then every 3 months till 6 months after the procedure
  Neck disability index (NDI, 35-point scale); 0-4points (0-8%) no disability, 5-14points (10 - 28%) mild disability, 15-24points (30-48% ) moderate disability, 25-34points (50- 64%) severe disability, 35-50points (70-100%) complete disability
Level of patient satisfaction | pre-procedure then every 3 months till 6 months after the procedure
  Level of patient satisfaction (5-point scale); Very dissatisfied Dissatisfied Neutral Satisfied Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Enas A Abd el Motlb, MD, Study Chair — Associate Professor
Locations (1):
- Enas A Abd el Motlb, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided